CLINICAL TRIAL: NCT05448287
Title: Suaahara Impact Evaluation: End-line Survey
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Helen Keller International (Other)
Responsible Party: Principal Investigator, Edward Frongillo, Jr., Professor, University of South Carolina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 103
Record Dates: First submitted 2022-06-16; First posted 2022-07-07 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Nutritional Stunting; Feeding Behavior
MeSH Terms: conditions — Feeding Behavior | interventions — Health; Family Planning Services; Nutritional Status; Agriculture; Water; Sanitation; Hygiene

STUDY DESIGN:
Intervention Model Description: Two-arm quasi-experimental design with baseline and end-line. The baseline and end-line were collected on different households but in the same clusters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Suaahara interventions span health and family planning; nutrition; agriculture/homestead food production; and water, sanitation and hygiene (WASH). Diverse social and behavior change communication interventions are used, primarily to generate demand for access to improved services and to motivate households to adopt optimal health, nutrition, and WASH practices. All Suaahara interventions are supported by a crosscutting theme of gender equality and social inclusion (GESI), in part by targeting women and disadvantaged groups and conducting activities that address GESI-related barriers to optimal health, nutrition, and WASH behaviors.
  Interventions: Behavioral: Health and family planning; Behavioral: Nutrition; Behavioral: Agriculture and homestead food production; Behavioral: Water, sanitation, and hygiene
- Comparison (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Health and family planning — Promotion of health and family planning behaviors
  Arms: Intervention
Behavioral: Nutrition — Promotion of maternal, infant, and young child feeding behaviors and nutrition
  Arms: Intervention
Behavioral: Agriculture and homestead food production — Promotion of knowledge and practices about homestead food production
  Arms: Intervention
Behavioral: Water, sanitation, and hygiene — Promotion of behaviors to improve water, sanitation, and hygiene
  Arms: Intervention

SUMMARY:
Suaahara's primary aim is to reduce the prevalence of stunting, wasting, and underweight among children under 5 years of age and to reduce the prevalence of anemia among women of reproductive age and children 6-59 months of age. For this, the program uses a multi-sectoral approach to achieve four key intermediate results: 1) improved household nutrition, sanitation, and health behaviors; 2) increased use of quality nutrition and health services by women and children; 3) improved access to diverse and nutrient-rich foods by women and children; and 4) accelerated roll-out of the Multi-Sectoral Nutrition Plan (MSNP) through strengthened local governance

DETAILED DESCRIPTION:
The Government of Nepal and development partners have prioritized multi-sectoral (integrated) nutrition as a key development agenda. The Suaahara program funded by the United States Agency for International Development is one of the programs that support the Government of Nepal's multi-sectoral nutrition plan. It aims to reduce maternal and child under-nutrition over a period of ten years, spanning two phases: Suaahara I (2011-2016) and Suaahara II (2016-2021). Initially launched in 20 of 75 districts, the program has scaled-up to 42 of 77 districts that span across Nepal's three agroecological zones of mountains, hills, and terai.

Suaahara I was led by Save the Children International in partnership with Helen Keller International, Johns Hopkins University Center for Communications Programs, Jhpiego, Nepal Water for Health (NEWAH), the National Promotion and Consultancy Service, and the Nepali Technical Assistance Group (NTAG). Suaahara II was led by Helen Keller International in partnership with Cooperative for Assistance and Relief Everywhere, Inc., Family Health International 360), he Nepali Technical Assistance Group, Digital Broadcast Initiative Equal Access, Environmental and Public Health Organization, and Vijaya Development Resource Center.

Suaahara's primary aim is to reduce the prevalence of stunting, wasting, and underweight among children under 5 years of age and to reduce the prevalence of anemia among women of reproductive age and children 6-59 months of age. For this, the program uses a multi-sectoral approach to achieve four key intermediate results (IRs): 1) improved household nutrition, sanitation, and health behaviors; 2) increased use of quality nutrition and health services by women and children; 3) improved access to diverse and nutrient-rich foods by women and children; and 4) accelerated roll-out of the MSNP through strengthened local governance. Suaahara interventions span health and family planning (FP), nutrition, agriculture/homestead food production (HFP), and water, sanitation and hygiene (WASH). Diverse social and behavior change communication interventions are used, primarily to generate demand for access to improved services and to motivate households to adopt optimal health, nutrition, and WASH practices. All Suaahara interventions are supported by a crosscutting theme of gender equality and social inclusion (GESI), in part by targeting women and disadvantaged groups and conducting activities that address GESI-related barriers to optimal health, nutrition, and WASH behaviors. Suaahara's conceptual framework illustrates the paths by which the program activities linked to desired outcomes achieve Suaahara II objectives.

ELIGIBILITY:
Inclusion Criteria:

* At the household level, the primary respondents are mothers of children under 5 years of age from the selected households.
* Other survey respondents include a primary male (or female, if male unavailable) household decision-maker, and a grandmother of children under 5 years of age residing in the household.
* The Female Community Health Volunteer and health workers are also Suaahara beneficiaries, as the program explicitly aims to improve their knowledge and skills.

Exclusion Criteria:

* None.

Ages: 0 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2480 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Child dietary diversity (Indicators for Assessing Infant and Young Child Feeding Practices) | Over the 24 hours of the day before data collection
  Mean score, range 0 to 8, higher is better
Maternal dietary diversity (Minimum Dietary Diversity for Women) | Over the 24 hours of the day before data collection
  Mean score, range 0 to 10, higher is better
Stunting | Over the 24 hours of the day of data collection
  Prevalence of height or length for age zscore < -2
Underweight prevalence | Over the 24 hours of the day of data collection
  Prevalence of weight for age zscore < -2
Wasting | Over the 24 hours of the day of data collection
  Prevalence of weight for length for height zscore < -2
Maternal underweight | Over the 24 hours of the day of data collection
  Prevalence of body mass index < 18.5
Maternal anemia | Over the 24 hours of the day of data collection
  Prevalence < 12 g/dl
Anemia among children aged 6-59 months | Over the 24 hours of the day of data collection
  Prevalence < 11 g/dl
Accurate health, nutrition, and water, sanitation, and hygiene knowledge and skills among Female Community Health Volunteers and health workers from 52 items | Over the 24 hours of the day of data collection
  Prevalence > 80% correct from 52 items

SECONDARY OUTCOMES:
Child minimum dietary diversity (Indicators for Assessing Infant and Young Child Feeding Practices) | Over the 24 hours of the day before data collection
  Prevalence > 4 food groups of 8
Maternal minimum dietary diversity (Minimum Dietary Diversity for Women) | Over the 24 hours of the day before data collection
  Prevalence > 4 food groups of 10
Height for age | Over the 24 hours of the day of data collection
  Mean z-score
Weight for age | Over the 24 hours of the day of data collection
  Mean z-score
Weight for height | Over the 24 hours of the day of data collection
  Mean z-score
Maternal body mass index | Over the 24 hours of the day of data collection
  Mean
Maternal hemoglobin | Over the 24 hours of the day of data collection
  Mean in g/dl
Child hemoglobin | Over the 24 hours of the day of data collection
  Mean in g/dl
Knowledge score on core infant and young child feeding practices among mothers from 15 items | Over the 24 hours of the day of data collection
  Mean score, range 0 to 15, higher is better
Knowledge score on health and water, sanitation, and hygiene practices among mothers from 37 items | Over the 24 hours of the day of data collection
  Mean score, range 0 to 37, higher is better
Female Community Health Volunteers and health workers with ideal practices related to health, nutrition, and water, sanitation, and health from 52 items | Over the 24 hours of the day of data collection
  Prevalence > 80% correct from 52 items

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Frongillo, PhD, Principal Investigator — University of South Carolina
Locations (1):
- Helen Keller International, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frongillo EA, Suresh S, Thapa DK, Cunningham K, Pandey Rana P, Adhikari RP, Kole S, Pun B, Kshetri I, Adhikari DP, Klemm R. Impact of Suaahara, an integrated nutrition programme, on maternal and child nutrition at scale in Nepal. Matern Child Nutr. 2026 Mar;22(1):e13630. doi: 10.1111/mcn.13630. Epub 2024 Feb 11. PMID 38342986